CLINICAL TRIAL: NCT04157192
Title: Brain Connectome for Migraine Patients Treated Via Acupuncture: A Randomized, Controlled Study Under Single-blind Conditions, With a Placebo Group and Magnetic Resonance Imaging (MRI)
Brief Title: Brain Connectome for Acupuncture-treated Migraine Patients
Acronym: ACU-BRAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCB : 2019-A00588-49
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Migraine Without Aura; Acupuncture Therapy
Keywords: Acupuncture
MeSH Terms: conditions — Migraine without Aura

STUDY DESIGN:
Intervention Model Description: 40 patients will be randomly assigned to one of two groups (1) The Interventional Group: 20 Patients will receive 5 real acupuncture sessions each spaced 15 days apart. At the first and last sessions of acupuncture, an MRI scan will be performed before and after the acupuncture session and (2) The Placebo Group : 20 patients will receive 5 sham sessions of acupuncture (i.e. using a simulated acupuncture technique) each spaced 15 days apart. At the first and last sham sessions, an MRI scan will be performed before and after the sham acupuncture session.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient is unaware of the study (and whether he/she is receiving the placebo or not).
  The imager is also unaware of whether the patient has had sham or real acupuncture.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients receiving real acupuncture treatment (Active Comparator): Treatment with needle insertion
  Interventions: Other: Real acupuncture
- Patients receiving sham acupuncture treatment (Sham Comparator): Treatment without needle insertion
  Interventions: Other: Sham acupuncture (placebo group)

INTERVENTIONS:
Other: Real acupuncture — The patient will be treated for migraine with real acupuncture.
  Arms: Patients receiving real acupuncture treatment
Other: Sham acupuncture (placebo group) — Sham acupuncture is used as a control in scientific studies to test the efficacy of acupuncture in the treatment of various disorders, in this case, migraine. In this study, the subjects will not know whether they are getting true acupuncture or not. In the placebo group, the acupuncture needles will not actually be inserted into the skin. Placebo needles consisting of a sliding tube and a retractible needle are applied to the acupunture reference point (marked by a pastille stuck on the skin). The patient should not be able to feel the difference between real acupuncture and sham acupuncture.
  Arms: Patients receiving sham acupuncture treatment

SUMMARY:
Acupuncture has been a means of treating headaches and migraine since 2002 and is now a World Health Organisation-recognized prophylactic treatment for migraine. Brain activation/de-activation via acupuncture modifies the haemodynamic responses in the brain which may impact the sensorial, cognitive and affective dimensions of pain. Randomized studies on patients suffering from aura-free migraine have shown that the painkilling effect of regular acupuncture sessions on the cerebral substratum, compared with simulated sham-type acupuncture, can reduce the frequency of bouts of migraine, number of days with headaches and also their intensity.

Modifications to the white matter (WM) and grey matter (GM) occur after repeated sessions of acupuncture treatment for pain and these are observable via magnetic resonance imaging (MRI). It is a very sensitive technique and often used to detect functional and structural brain changes.

DETAILED DESCRIPTION:
Since 2002, acupuncture has been employed as a method for treating headaches and migraine. It is recognized by the World Health Organisation (WHO), and is now part of the prophylactic treatments for migraine. Brain activations/de-activation via acupuncture lead to a modification of haemodynamic responses in the brain which may impact the sensorial, cognitive and affective dimensions of pain. Randomized studies on patients who suffer from migraine without aura have shown that the painkilling effect of repeated acupuncture sessions on the cerebral substratum, compared with simulated sham-type acupuncture, make it possible to reduce the frequency of bouts of migraine, the number of days of headaches, and the intensity of the bouts.

Following repeated sessions of acupuncture treatment for pain, modifications occur in the white matter (WM) and in the grey matter (GM) and these may be observed by magnetic resonance imaging (MRI) which is a highly sensitive technique and very often used to detect functional brain changes and/or subtle abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* All patients with two to eight bouts of migraine without an aura per month
* All patient aged (≥) 18 to (≤) 60 years old
* All patients who have not had a bout of migraine in the last 24 hours
* All patients who have given free informed consent and have signed the consent form.
* All patients who are affiliated to or beneficiaries of a health insurance scheme
* All patients available for a two-month follow-up

Exclusion Criteria:

* All patients with migraine which is secondary to a neurological, neuropsychiatric, or vascular disorder
* All patients suffering from diabetes
* All patients with a past history of alcohol or drug abuse
* All patients with contraindications for an MRI scan
* All patients on antidepressants or Botox.
* All patients already taking part in Category 1 research involving the human person
* All patients on an exclusion period determined by another study
* All patients placed under judicial protection, guardianship, or supervision
* All patients for whom it is impossible to give the subject clear information
* All patients who are pregnant, about to give birth or breastfeeding
* All patient who have received botulinum toxin in the past year
* All patient who have undergone antidepressant treatment in the last 2 months
* All patient who have started a background migraine treatment for less than 3 months
* All patient who have more than 14 migraine days per month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Regional homogeneity map in Interventional group patients BEFORE first real acupuncture session. | At the inclusion visit (Vinc) on Day 0 - Start of therapy
  Regional homogeneity in patients treated via real acupuncture (Interventional group) is computed with functional magnetic resonance imaging
Regional homogeneity map in Interventional group patients AFTER first real acupuncture session. | At the inclusion visit (Vinc) on Day 0 - Start of therapy
  Regional homogeneity in patients treated via real acupuncture (Interventional group) is computed with functional magnetic resonance imaging
Regional homogeneity map in Placebo group patients BEFORE first real acupuncture session. | At the inclusion visit (Vinc) on Day 0 - Start of therapy
  Regional homogeneity in patients treated via simulated, sham-type acupuncture (Placebo group) is computed with functional magnetic resonance imaging
Regional homogeneity map in Placebo group patients AFTER first real acupuncture session. | At the inclusion visit (Vinc) on Day 0 - Start of therapy
  Regional homogeneity in patients treated via simulated, sham-type acupuncture (Placebo group) is computed with functional magnetic resonance imaging
Regional homogeneity map in Interventional group patients BEFORE last real acupuncure session | Sixty days after inclusion in the trial (Day 60) - end of therapy
  Regional homogeneity in patients treated via acupuncture (Interventional group) is is computed with functional magnetic resonance imaging
Regional homogeneity map in Interventional group patients AFTER last real acupuncure session | Sixty days after inclusion in the trial (Day 60) - end of therapy
  Regional homogeneity in patients treated via acupuncture (Interventional group) is computed with functional magnetic resonance imaging
Regional homogeneity map of Placebo group patients BEFORE last placebo acupuncture session | Sixty days after inclusion in the trial (Day 60) - end of therapy
  Regional homogeneity in patients treated via simulated, sham-type acupuncture (Placebo group) is computed with functional magnetic resonance imaging
Regional homogeneity map of Placebo group patients AFTER last placebo acupuncture session | Sixty days after inclusion in the trial (Day 60) - end of therapy
  Regional homogeneity in patients treated via simulated, sham-type acupuncture (Placebo group) is computed with functional magnetic resonance imaging

SECONDARY OUTCOMES:
Mean diffusivity of White Matter of Interventional group patients BEFORE first real acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  The mean diffusivity of White Matter of Interventional group patients is computed with diffusion-weighted magnetic resonance imaging
Mean diffusivity of White Matter of Interventional group patients AFTER first real acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  The mean diffusivity of White Matter of Interventional group patients is computed with diffusion-weighted magnetic resonance imaging
Mean diffusivity of White Matter of Placebo group patients BEFORE first placebo acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  The mean diffusivity of White Matter of Placebo group patients is computed with diffusion-weighted magnetic resonance imaging
Mean diffusivity of White Matter of Placebo group patients AFTER first placebo acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  The mean diffusivity of White Matter of Placebo group patients is computed with diffusion-weighted magnetic resonance imaging
Mean diffusivity of White Matter of Interventional group patients BEFORE last real acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  The mean diffusivity of White Matter in patients treated with real acupuncture (Interventional group) is computed with diffusion-weighted magnetic resonance imaging
Mean diffusivity of White Matter of Interventional group patients AFTER last real acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  The mean diffusivity of White Matter in patients treated with real acupuncture (Interventional group) is computed with diffusion-weighted magnetic resonance imaging
Mean diffusivity of White Matter of Placebo group patients BEFORE last placebo acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  The mean diffusivity of White Matter in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Mean diffusivity of White Matter of Placebo group patients AFTER last placebo acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  The mean diffusivity of White Matter in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Radial diffusivity of the White Matter in Interventional group patients BEFORE first real acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  Radial diffusivity of the White Matter of Interventional group patients is computed with diffusion-weighted magnetic resonance imaging
Radial diffusivity of the White Matter in Interventional group patients AFTER first real acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  Radial diffusivity of the White Matter in the Interventional group patients is computed with diffusion-weighted magnetic resonance imaging
Radial diffusivity of the White Matter in Placebo group patients BEFORE first placebo acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  Radial diffusivity of the White Matter in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Radial diffusivity of the White Matter in Placebo group patients AFTER first placebo acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  Radial diffusivity of the White Matter in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Radial diffusivity of the White Matter in Interventional group patients BEFORE last real acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  Radial diffusivity of the White Matter in patients treated with real acupuncture (Interventional group) is computed with diffusion-weighted magnetic resonance imaging
Radial diffusivity of the White Matter in Placebo group patients AFTER last real acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  Radial diffusivity of the White Matter in patients treated with real acupuncture (Interventional group) is computed with diffusion-weighted magnetic resonance imaging
Radial diffusivity of the White Matter in Interventional group patients BEFORE last placebo acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  Radial diffusivity of the White Matter in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Radial diffusivity of the White Matter in Placebo group patients AFTER last placebo acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  Radial diffusivity of the White Matter in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Fractional anisotropy of the White Matter in Interventional group patients BEFORE first real acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  Fractional anisotropy of patients treated with real acupuncture (Interventional group) is computed with diffusion-weighted magnetic resonance imaging
Fractional anisotropy of the White Matter in Interventional group patients AFTER first real acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  Fractional anisotropy of patients treated with real acupuncture (Interventional group) is computed with diffusion-weighted magnetic resonance imaging
Fractional anisotropy of the White Matter in Placebo group patients BEFORE first placebo acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  Fractional anisotropy in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Fractional anisotropy of the White Matter in Placebo group patients AFTER first placebo acupuncture session | At the inclusion visit (Vinc) on Day 0 - start of therapy
  Fractional anisotropy in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Fractional anisotropy of the White Matter in Interventional group patients BEFORE last real acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  Fractional anisotropy in patients treated with real acupuncture (Interventional group) is computed with diffusion-weighted magnetic resonance imaging
Fractional anisotropy of the White Matter in Interventional group patients AFTER last real acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  Fractional anisotropy in patients treated with real acupuncture (Interventional group) is computed with diffusion-weighted magnetic resonance imaging
Fractional anisotropy of the White Matter in Placebo group patients BEFORE last placebo acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  Fractional anisotropy in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Fractional anisotropy of the White Matter in Placebo group patients AFTER first placebo acupuncture session | 60 days after the initial inclusion visit (Day 60) - end of therapy
  Fractional anisotropy in patients treated with simulated, sham-type acupuncture (Placebo group) is computed with diffusion-weighted magnetic resonance imaging
Change in number of days with migraine per month - Interventional group BEFORE treatment | At the inclusion visit (Vinc) on Day 0
  The number of days with migraine per month will be measured according to the days noted on a calendar
Change in number of days with migraine per month - Interventional group AFTER treatment | At the end of the study (on Day 90)
  The number of days with migraine per month will be measured according to the days noted on a calendar
Change in number of days with migraine per month - Placebo group BEFORE treatment | At the inclusion visit (Vinc) on Day 0
  The number of days with migraine per month will be measured according to the days noted on a calendar
Change in number of days with migraine per month - Placebo group AFTER treatment | At the end of the study (on Day 90)
  The number of days with migraine per month will be measured according to the days noted on a calendar
Pain BEFORE treatment in the Interventional group | At the inclusion visit (Vinc) on Day 0
  The change in pain will be measured according to the Visual Analogue Scale (VAS) described by Huskisson. The VAS is a simple numerical scale for measuring the intensity of pain. It is represented in the form of a 100 mm continuous line ranging from "Absence of pain" (0 mm) to "Maximum Imaginable Pain" (100 mm). The patient slides the cursor to give the intensity of pain that he/she feels. The amount of pain felt will be reported on the migraine calendar.
Pain AFTER treatment in the Interventional group | At the end of the study (on Day 90)
  The change in pain will be measured according to the Visual Analogue Scale (VAS) described by Huskisson. The VAS is a simple numerical scale for measuring the intensity of pain. It is represented in the form of a 100 mm continuous line ranging from "Absence of pain" (0 mm) to "Maximum Imaginable Pain" (100 mm). The patient slides the cursor to give the intensity of pain that he/she feels. The amount of pain felt will be reported on the migraine calendar.
Pain BEFORE treatment in the Placebo group | At the inclusion visit (Vinc) on Day 0
  The change in pain will be measured according to the Visual Analogue Scale (VAS) described by Huskisson. The VAS is a simple numerical scale for measuring the intensity of pain. It is represented in the form of a 100 mm continuous line ranging from "Absence of pain" (0 mm) to "Maximum Imaginable Pain" (100 mm). The patient slides the cursor to give the intensity of pain that he/she feels. The amount of pain felt will be reported on the migraine calendar.
Pain AFTER treatment in the Placebo group | At the end of the study (on Day 90)
  The change in pain will be measured according to the Visual Analogue Scale (VAS) described by Huskisson. The VAS is a simple numerical scale for measuring the intensity of pain. It is represented in the form of a 100 mm continuous line ranging from "Absence of pain" (0 mm) to "Maximum Imaginable Pain" (100 mm). The patient slides the cursor to give the intensity of pain that he/she feels. The amount of pain felt will be reported on the migraine calendar.
Impact of migraine on the Interventional group patients' Quality of Life (QOL) BEFORE treatment | At the inclusion visit (Vinc) on Day 0
  The evolution of the impact of migraine on the patient's Quality of Life (QOL) before and after treatment will be measured on a score of 36 to 78 points by means of the Headache Impact Test-6 (HIT-6). This is a tool used to measure the impact of headaches on the patient's ability to function at work, at school, at home and in social situations.
Impact of migraine on the Interventional group patients' Quality of Life (QOL) AFTER treatment | At the end of the study on Day 90
  The evolution of the impact of migraine on the patient's Quality of Life (QOL) before and after treatment will be measured on a score of 36 to 78 points by means of the Headache Impact Test-6 (HIT-6). This is a tool used to measure the impact of headaches on the patient's ability to function at work, at school, at home and in social situations.
Impact of migraine on the Placebo group patients' Quality of Life (QOL) BEFORE treatment. | At the inclusion visit (Vinc) on Day 0
  The evolution of the impact of migraine on the patient's Quality of Life (QOL) before and after treatment will be measured on a score of 36 to 78 points by means of the Headache Impact Test-6 (HIT-6). This is a tool used to measure the impact of headaches on the patient's ability to function at work, at school, at home and in social situations.
Impact of migraine on the Placebo group patients' Quality of Life (QOL) AFTER treatment. | At the end of the study on Day 90
  The evolution of the impact of migraine on the patient's Quality of Life (QOL) before and after treatment will be measured on a score of 36 to 78 points by means of the Headache Impact Test-6 (HIT-6). This is a tool used to measure the impact of headaches on the patient's ability to function at work, at school, at home and in social situations.

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Mme., Study Director — CHU de Nîmes (Nîmes University Hospital)
Locations (1):
- Marc FREARD, Nîmes, France